CLINICAL TRIAL: NCT00138034
Title: A Multicenter Randomized Trial in the Prevention of Reocclusion Following Successful Thrombolysis for Suspected Acute Myocardial Infarction: An Invasive Versus a Conservative Strategy
Brief Title: APRICOT-3: Antithrombotics in the Prevention of Reocclusion In COronary Thrombolysis -3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heartcenter, University Medical Center St. Radboud (Other)
Collaborators: Netherlands Heart Foundation (Other); The Interuniversity Cardiology Institute of the Netherlands (Other Government); Pfizer (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Prof. Dr. F.W.A. Verheugt, Professor of Cardiology, Heartcenter, University Medical Center St. Radboud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APRICOT-3; 2003B257 (Other: Netherlands Heart Foundation)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Myocardial Infarction
Keywords: Open infarct-related artery within 72 hours of thrombolysis
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous coronary intervention (PCI) (Active Comparator): Stenting of the culprit lesion of the infarct related artery and aspirin and clopidorgel for at least 6 months
  Interventions: Procedure: Percutaneous coronary intervention (PCI)
- Dual antiplatelet therapy (Other): Aspirin and clopidogrel for at least 6 months
  Interventions: Procedure: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — PCI with bare metal stent placement of the culprit lesion the in the infarct related artery
  Other Names: bare metal stent placement

SUMMARY:
Reocclusion of the infarct artery is observed in about 30% of patients within three months after successful thrombolysis for acute myocardial infarction (MI). Reocclusion is associated with an increased risk of death, reinfarction and the need for revascularization. Even in the absence of clinical reinfarction, reocclusion results in impaired left ventricular (LV) recovery, leaving patients at increased risk of developing heart failure in the long-term. Prevention of reocclusion is therefore warranted. In previous trials, severity of the infarct related stenosis was the only independent predictor of reocclusion. With a lack of clinical predictors of reocclusion, many cardiologists therefore empirically favor routine revascularization after successful thrombolysis.

The APRICOT-3 will be the first randomized trial in the current era of improved angioplasty techniques to study the question of whether a routine invasive strategy after successful thrombolysis can reduce the incidence of reocclusion and subsequently improve clinical outcome and LV-function. After successful thrombolysis, patients will be randomized to either a routine invasive strategy or an ischemia-guided strategy. The investigators expect to demonstrate a lower reocclusion rate at the 6-month follow-up angiography (primary endpoint) and fewer associated events (death, reinfarction, revascularization, admissions for heart failure) in the routine invasive arm. In search of non-invasive parameters predictive of reocclusion, laboratory analysis of several coagulation and inflammatory markers will be performed. Finally, pooled analysis of all 3 APRICOT trials will focus on the identification of clinical predictors of reocclusion that can easily be obtained by history and physical examination.

DETAILED DESCRIPTION:
Randomized controlled study of elective percutaneous coronary intervention (PCI) of an open culprit lesion after fibrinolysis for ST-elevation myocardial infarction (STEMI)

ELIGIBILITY:
Inclusion Criteria:

* TIMI-3 in infarct-related artery with a stentable lesion with 72 hours of thrombolysis for ST-elevation myocardial infarction

Exclusion Criteria:

* Use of oral anticoagulants.
* Known intolerance to aspirin or clopidogrel.
* Bypass graft as infarct-related artery.
* Previously dilated infarct related artery.
* Significant left main stenosis.
* Unidentifiable culprit stenosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-01; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Freek WA Verheugt, MD PhD, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were included from 1 january 2005 until december 2009
Groups:
- Percutaeous Coronary Intervention (PCI): Stenting of culprit lesion followed by dual antiplatelet therapy
- Conservative Treatment: Conservative treatment of culprit lesion with dual antiplatelet therapy
Period: Overall Study
Arm/Group | Percutaeous Coronary Intervention (PCI) | Conservative Treatment
Started | 26 | 23
Completed | 23 | 20
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaeous Coronary Intervention (PCI) | Conservative Treatment | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 10 | 8 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 59 (13) | 59 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 22 | 19 | 41
Region of Enrollment [Number; unit: participants]
  Netherlands | 20 | 20 | 40
  Austria | 2 | 1 | 3
  Australia | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: 6-month Reocclusion
Description: Less than TIMI (Thrombolysis In Myocardial Infarction) -3 flow of the infarct related coronary artery assessed at follow-up angiography
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Percutaeous Coronary Intervention (PCI) | Conservative Treatment
Number analyzed (Participants) | 26 | 23
participants | 1 | 4

2. Secondary Outcome: Composite of Death, Reinfarction, Stroke and Revascularization at the Time of Follow-up Angiography
Description: The occurence of any one of the above mentioned outcome measures. Only the first event per patient is counted.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Percutaeous Coronary Intervention (PCI) | Conservative Treatment
Number analyzed (Participants) | 26 | 23
participants | 4 | 7

ADVERSE EVENTS:
Arm/Group | Percutaeous Coronary Intervention (PCI) | Conservative Treatment
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaeous Coronary Intervention (PCI) (N=26) | Conservative Treatment (N=23)
intracerebral bleeding (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Freek W.A. Verheugt

has to following potential conflict of interest:

1. received educational and research grants from Bayer Healthcare, Roche, Eli Lilly and Boehringer Ingelheim
2. received honoraria for consultancies from Daiichi-Sankyo, Eli Lilly, Merck, The Medicines Company and Bayer Healthcare